CLINICAL TRIAL: NCT00729235
Title: Biventricular Tachycardias Outcome Trial
Acronym: BITAC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: LivaNova (Industry)
Responsible Party: Alexander Bauer / Principal investigator, Universitätsklinikum Heidelberg
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BITAC - ITAC04
Record Dates: First submitted 2008-08-04; First posted 2008-08-07 (Estimated); Last update posted 2011-12-22 (Estimated); Status verified 2010-06

CONDITIONS: Biventricular Tachycardias
Keywords: Slow VT, CRT-D, ATP therapy; Incidence; of slow VTs; in CRT-D patients; Clinical; relevance; treatment; VTs; during; 2-years; follow-up

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Slow VT zone programmed as a "Monitoring" zone (Monitoring arm)
  Interventions: Device: Ovatio CRT 6750
- 2 (Experimental): Slow VT zone programmed with ATP therapies (therapy arm).
  Interventions: Device: Ovatio CRT 6750

INTERVENTIONS:
Device: Ovatio CRT 6750 — Slow VT zone programmed as a "Monitoring" zone (Monitoring arm)
  Arms: 1
Device: Ovatio CRT 6750 — Slow VT zone programmed with ATP therapies (therapy arm).
  Arms: 2

SUMMARY:
This clinical investigation is a device-based open, prospective, multicenter two-arm randomized trial, comparing patients who are treated in the slow VT zone versus patients who are not treated in that zone.

The device intended to be used is the OVATIOTM CRT model 6750 but future generation of Sorin Group/ ELA Medical devices may be used provided they are CE marked. Ethics committees and health authorities will be informed prior to any use of a newer device if applicable.

All patients will have a 3-zone detection configuration programmed. The slow VT zone will be defined by programming the detection parameters as follows:

* Slow VT detection rate: 100 bpm (or if the resting rate is higher than 80 bpm, we recommend to adjust this parameter to: resting rate + 30 bpm)
* VT detection rate: 150 bpm

PARAD+ will be the first choice for SVT/ST and VT discrimination in the VT zones.

The Fast VT and VF limits are left to investigator's judgment. Therapy on VT, fast VT and VF are also left to the investigator's judgment.

Patients will be randomized at implant to have the slow VT zone programmed as a monitoring zone (monitoring arm) or to have therapies programmed within the slow VT zone (therapy arm). The randomization table will be generated by Sorin Group/ELA Medical.

ELIGIBILITY:
Inclusion Criteria:

* Patient has been prescribed the implantation or replacement of a CRT-ICD system accordingly to the relevant currently-approved ACC/AHA15 (August 2005, Appendix §M.10) or ESC 16 (Update 2005, Appendix § M.11) guidelines or any relevant currently-approved local guidelines for the implantation or replacement of CRT-ICD.
* Patient has signed a consent form after he/she received the appropriate and mandatory information.

Exclusion Criteria:

* Clinical history of symptomatic or not symptomatic slow VT;
* Permanent Atrial Fibrillation (AF);
* Any contraindication to the implant or replacement of CRT-ICD;
* Pt is unable to attend the scheduled f-up visits at the implanting Centre;
* Pt is already included in another ongoing clinical study;
* Pt is unable to understand the objectives of the ITAC04 study;
* Pt refuses to cooperate;
* Pt is unable or refuses to provide informed consent;
* Pt is minor (less than 18-year old);
* Pt has life expectancy of less than 1 year;
* Pt is pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 481 (Actual)
Dates: Start 2006-05; Primary Completion 2008-12 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Incidence of slow ventricular tachycardias (Slow VTs) in CRT-ICD pts; | 24 months
ATP therapy efficacy on slow VTs conversion. | 24 months

SECONDARY OUTCOMES:
Efficacy of ATP therapies on Slow VTs according to therapy setting (delivery in LV only, in RV only, or in LV+RV) | 24 months
Tvar risk stratification | 24 months
"unscheduled visits" or "hospital re-admissions" due to slow VTs; | 24 months
Incidence of adverse events (AEs) in the studied population | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Bauer, Principal Investigator — Universitätsklinikum Heidelberg, 69120 Heidelberg
Locations (49):
- Algemeen Ziekenhuis, Antwepen, Belgium
- Canada (3):
  - Grey-Nuns Hospital, Edmonton
  - Royal Alexandra Hospital, Edmonton
  - Laval UH, Ste Foy, Québec
- France (25):
  - CH Albi, Albi
  - CH Angers, Angers
  - Hôpital privé d'Antony, Antony
  - Hôpital Haut Lévèque, Bordeaux
  - Hôpital de la Cavalle Blanche, Brest
  - Clinique de Parly II, Le Chesnay
  - CH St Philibert, Lomme
  - CHU Hopital La Timone, Marseille
  - CHU Hôpital Nord - Marseille, Marseille
  - CHU Hôpital Nord, Marseille
  - Clinique Beauregard, Marseille
  - Clinique Clairval, Marseille
  - Hôpital Arnaud de Villeneu, Montpellier
  - Clinique Amboise Paré, Neuilly
  - CHU Hopital Pasteur, Nice
  - CHU Groupe Carémeau, Nîmes
  - C.H.R Hopital De La Source, Orléans
  - Clinique Bizet, Paris
  - CH Pau, Pau
  - Hôpital de la Miletrie, Poitiers
  - CHU Charles Nicolle, Rouen
  - Centre Cardiologique Du Nord, Saint-Denis
  - CHU Hôpital Nord, Saint-Etienne
  - Hopital Font Pré, Toulon
  - Hôpital Purpan, Toulouse
- Germany (8):
  - Herzkreislaufklinik, Bad Bevensen
  - Kerckhoff-Klinik GmbH, Bad Nauheim
  - Praxis Westend, Berlin
  - Universitatsklinik Med. Klinik Heidelberg, Heidelberg
  - Universität des Saarlandes, Homburg
  - Universitätsklinikum Schleswig-Holstein, Lübeck
  - Uniklinik Munster, Münster
  - Krankenhaus Reinbek, Reinbek
- Italy (3):
  - Ospedale Civile Di Asti, Asti
  - Casa di cura villa pini d'abruzo, Chieti
  - Hospital Clinico, Valencia
- Hospital Fernando Fonseca, Amadora, Portugal
- CHUVI, Vigo, Spain
- Sweden (2):
  - Danderyds Sjukhus Ab, Danderyd
  - Orebro Universitetssjukhus, Örebro
- United Kingdom (5):
  - Royal Bournemouth Hospital, Bournemouth
  - Glenfield Hospital, Leicester
  - St Barts Hospital, London
  - Northern General Hospital, Sheffield
  - Southampton General Hospital, Southampton